CLINICAL TRIAL: NCT05248334
Title: Ranibizumab in the Treatment of Postoperative Recurrent Vitreous Haemorrhage of Diabetic Retinopathy
Brief Title: A Prospective Study of Ranibizumab in the Treatment of Postoperative Recurrent Vitreous Haemorrhage of Diabetic Retinopathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Eye Hospital (Other)
Collaborators: Hebei Provincial Eye Hospital (Other); Cangzhou Eye Hospital (Unknown)
Responsible Party: Principal Investigator, Bojie Hu, Professor, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TianjinMUEHhbj123
Record Dates: First submitted 2022-02-07; First posted 2022-02-21 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Retinopathy; Postoperative Recurrent Vitreous Hemorrhage; Pars Plana Vitrectomy; Ranibizumab
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ranibizumab group (Experimental): The Ranibizumab group was treated with one intravitreal injection of 0.5 mg/0.05 ml ranibizumab (Lucentis, Basel, Novartis) at baseline. While additional panretinal photocoagulation was performed if there was sufficient space and view to fill in the previously untreated areas, if needed. Repeated injections will be given after 4 weeks when the clearing of VH was incomplete (for a maximum of two injections).
  If vitreous hemorrhage was not absorbed/vitreous hemorrhage aggravation/proliferation membrane formation/retinal detachment after 4 weeks of observation, the treatment was considered failed and PPV was performed.
  Interventions: Drug: Ranibizumab Injection
- PPV group (Active Comparator): Vitrectomy to remove vitreous hemorrhage and take additional panretinal photocoagulation. If vitreous hemorrhage was not absorbed/vitreous hemorrhage aggravation/proliferation membrane formation/tractive retinal detachment after 4 weeks of observation, the treatment was considered failed and PPV was performed.
  Interventions: Procedure: PPV

INTERVENTIONS:
Drug: Ranibizumab Injection — The Ranibizumab group was treated with one intravitreal injection of 0.5 mg/0.05 ml ranibizumab (Lucentis, Basel, Novartis) at baseline. While additional panretinal photocoagulation was performed if there was sufficient space and view to fill in the previously untreated areas, if needed. Repeated injections will be given after 4 weeks when the clearing of VH was incomplete (for a maximum of two injections).
  If vitreous hemorrhage was not absorbed/vitreous hemorrhage aggravation/proliferation membrane formation/retinal detachment after 4 weeks of observation, the treatment was considered failed and PPV was performed.
  Other Names: Panretinal photocoagulation
  Arms: Ranibizumab group
Procedure: PPV — Vitrectomy to remove vitreous hemorrhage and take additional panretinal photocoagulation. If vitreous hemorrhage was not absorbed/vitreous hemorrhage aggravation/proliferation membrane formation/tractive retinal detachment after 4 weeks of observation, the treatment was considered failed and PPV was performed.
  Other Names: Panretinal photocoagulation
  Arms: PPV group

SUMMARY:
Diabetic retinopathy (DR) is one of the main complications in diabetes, the proliferative diabetic retinopathy (PDR) is the most important one of the reasons leading to decreased vision, PDR is the stage of clinical intervention. Pars plana vitrectomy (PPV) is an effective treatment for PDR, while vitreous haemorrhage (VH) is a common complication after PPV, with incidence ranging from 11.8% to 75%, and is the main cause of reoperation. Anti-Vascular endothelial growth factor (VEGF) therapy for vitreous hemorrhage can inhibit neovascularization and prevent recurrent vitreous haemorrhage after absorption. Previous studies have found that anti-VEGF is a safe and effective treatment for postoperative recurrent VH. In consideration of the psychological and economic factor of patients, this study intends to observe the effectiveness of single vitreous injection of Ranibizumab in the treatment of postoperative recurrent VH on the basis of previous clinical work. Compare the visual acuity, macular thickness, VH recurrence and patient satisfaction between the Ranibizumab group and the PPV group by randomized grouping.To observe the effective rate and clearance time of recurrent VH after Ranibizumab treatment and whether it can effectively reduce the rate of PPV. To provide clinical guidance for the precise treatment of PDR patients, the treatment of PDR patients has important clinical significance and social and economic significance.

DETAILED DESCRIPTION:
1. Patients with proliferative diabetic retinopathy who underwent vitrectomy were collected. Vitreous hemorrhage was completely cleared for more than 1 week after surgery, and vitreous recurrent hemorrhage was not absorbed for more than 4 weeks (grade 2 and above). If the patient has recurrent vitreous hemorrhage or symptoms suggestive of recurrent vitreous hemorrhage, ultrasound at 10mhz posterior segment and 20mhz anterior segment are performed by an experienced sonographer. Patients were randomly assigned to PPV group or Ranibizumab group according to the order in which they came to visit and according to a random number table.
2. PPV group: PPV and pan retinal photocoagulation; in the Ranibizumab group, Ranibizumab was injected and pan retinal photocoagulation was performed during ocular fundus could observed, and observation for 4 weeks. If vitreous hemorrhage was not absorbed/vitreous hemorrhage aggravation/proliferation membrane formation/ retinal detachment, PPV was performed.
3. Collected information: best corrected visual acuity, slit lamp and fundus examination, intraocular pressure, B-ultrasound, macular thickness, the date of recurrent vitreous hemorrhage and treatment, vitreous cleaning time, the time of significant improvement of visual acuity, times and duration of vitreous hemorrhage. The follow-up time was 1 day, 2 weeks, 1 month, 2 months, 4 months and 6 months, respectively. To observe the effectiveness of Ranibizumab in the treatment of postoperative recurrent vitreous hemorrhage and reduce the number of vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and able to sign an informed consent form
* Age ≥18 years
* Documented diagnosis of diabetes mellitus (type I or type II diabetes) as defined by the American Diabetes Association or World Health Organization criteria and glycosylated hemoglobin ≤10% within 2 months
* Willing and able to complete all planned visits and evaluations
* Complete Panretinal photocoagulation
* Retinal repositioning
* Complete postoperative vitreous hemorrhage clearance for more than 1 week and non-absorption of recurrent vitreous hemorrhage for more than 4 weeks (grade 2 and above)
* Early postoperative period (1 week to 1 month postoperatively) and delayed postoperative period (4 weeks to 12 months postoperatively)

Exclusion Criteria:

* Patients with less than 6 months of follow-up
* Silicone oil filling
* Other retinal causes of vitreous hemorrhage
* Tractive retinal detachment, pre-retinal proliferative membrane
* Iris redness, neovascular glaucoma
* History of glaucoma
* Ocular inflammation
* Any other intraocular surgery (e.g., corneal transplantation, glaucoma filtration, corneal transplantation therapy, etc.)
* Patients with best corrected visual acuity manual or worse, patients with a single eye
* Previous cerebrovascular or thromboembolic events, hypertensive disorders, renal disease, current use of anticoagulants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The cleaning time of postoperative recurrent vitreous hemorrhage | two months
  Record VH by B scan and funds examination
Visual acuity | six moths
  ETDRS Alphabet Chart

SECONDARY OUTCOMES:
Macular thickness | six moths
  optical coherence tomography (OCT); TOPCON 3D-OCT-2000; Topcon Corporation, Tokyo, Japan
Vitreous hemorrhage recurrence | six moths
  B scan and funds examination
The number of pars plana vitrectomy | six moths
  Record the number of pars plana vitrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China